CLINICAL TRIAL: NCT06712043
Title: Testing a Tailored Home Exercise Program to Gain Insight Into Performance Fatigability and Reduce Pain and Fatigue in Patients with FSHD: the GRIP on FSHD Study
Brief Title: Testing a Tailored Home Exercise Program to Reduce Pain and Fatigue in Patients with FSHD.
Acronym: GRIPonFSHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Università di Pavia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL86789.091.24
Record Dates: First submitted 2024-08-13; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: FSHD
Keywords: Personalized exercise; Rehabilitation; Aerobic exercise; Strength training; Balance training; Fatigue; Pain; Fatigability; Smartphone application
MeSH Terms: conditions — Fatigue; Pain

STUDY DESIGN:
Intervention Model Description: Single group intervention study with historical control group
Masking Description: Not possible in this situation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): An individualized exercise program consisting of aerobic exercises, strength exercises and balance exercises. The exercises will be prescribed via the Physitrack app.
  Interventions: Behavioral: Personalised Exercise
- Historical control group (Active Comparator): Aerobic training (see study Voet 2024, Both aerobic exercise and cognitive-behavioral therapy reduce chronic fatigue in FSHD)
  Interventions: Behavioral: Historical control group

INTERVENTIONS:
Behavioral: Personalised Exercise — An individualized exercise program consisting of aerobic exercises, strength exercises and balance exercises. The exercises will be prescribed via the Physitrack app.
  Arms: Intervention group
Behavioral: Historical control group — Aerobic training (see study Voet 2024, Both aerobic exercise and cognitive-behavioral therapy reduce chronic fatigue in FSHD)
  Arms: Historical control group

SUMMARY:
The goal of this intervention study is to determine the effect of a tailored exercise program (with aerobic, strength and balance training) in patients with FSHD.

The main aim is to determine the effect of the exercise program on pain and fatigue.

Participants will follow a 16 week training program with tailored exercises. The exercises will be prescribed via the app 'Physitrack'. After 16 weeks, the effect on pain, fatigue, fatigability, aerobic capacity, balance, physical function, sleep and the ability to participate in social activities will be determined.

DETAILED DESCRIPTION:
Rationale: Pain and fatigue are two common and disabling symptoms in FSHD. No studies in FSHD have proven to reduce pain yet. (Aerobic) exercise has proven to reduce fatigue, however, current training guidelines are generic which can lead to overuse of injuries. The investigators expect that a personalized training program with aerobic exercise but also strength and balance training, that is adapted to a participants symptoms and wishes will provide a positive effect on pain and fatigue.

Objectives:

Primary objectives

1. To determine the effect of a tailored exercise program by using the widely implemented exercise app "Physitrack" on experienced pain and fatigue in patients with FSHD.
2. To investigate the relationship between perceived pain and fatigue and performance fatigability, disease severity, clinical phenotype, and level of activity in patients with FSHD Secondary objectives

1. To determine the responsiveness of the performance fatigability test. 2. To investigate the influence of a decreasing performance fatigability on experienced fatigue 3. To provide input for new training guidelines for people with FSHD. Study design: Single group intervention study with historical control group. Study population: 50 individuals with FSHD >18 years Intervention: An individualized exercise program consisting of aerobic exercises, strength exercises and balance exercises. The exercises will be prescribed via the Physitrack app.

Main study parameters/endpoints:

The chronic fatigue score assessed using the Checklist Individual Strength (CIS-fatigue) fatigue subscale and the average daily pain score during 2 weeks are the primary endpoints.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participating in this study includes: (1) two visits to the Radboudumc (approximately 3-4 hours, including a break) with physical test and questionnaires, (2) following a 16 week personalized exercise program, including filling in questionnaires about pain and fatigue and (3) wearing an activity tracker for 1 week before and after the study. Participants will have a weekly phone call with the researcher, and when participants will have complaints such as pain and/or fatigue, the training will be adapted. Therefore, the investigators expect that the risk will be minimal, and patient might experience the benefits of personalized training.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Verified diagnosis of FSHD type 1, based on the clinical criteria established by Padberg et al. (1991) (22).
* Category A or B of the four clinical categories according to the Comprehensive Clinical Evaluation Form (23), these patients have the most peculiar signs of the disease
* A CIS-fatigue score of ≥ 35
* Owning of and being able to use a smartphone
* Preserved ability to ambulate at the time of the selection
* No pulmonary or cardiological involvement, that could interfere with physical training.
* Absence of central or peripheral nervous system involvement as from neurological history and physical assessment
* Absence of limb contractures and tendon retractions

Exclusion Criteria:

* Use of beta-blocker medication
* Presence of additional diseases likely to interfere with the measurements
* Psychological-psychiatric disorders
* A musculoskeletal injury that impairs exercising
* Scoliosis that impairs training
* Recent adjustment of any medications or medications that may impact fatigue or taking stimulants for fatigue (e.g., Modafinil, amantadine)
* Current participation in another clinical investigation of a medical device or a drug; or has participated in such a study within 30 days prior to this study
* Pregnant women
* Patient incapable of understanding the purpose and conditions of the study, incapable of giving consent or using the app
* Patient deprived of liberty or patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Daily observed pain | 16 weeks
  Daily observed pain during a period of 2 weeks, measured with the Visual Analog Scale (VAS)
Fatigue | 16 weeks
  The chronic fatigue score assessed using the Checklist Individual Strength (CIS-fatigue) fatigue subscale.

SECONDARY OUTCOMES:
Performance fatigability | 16 weeks
  The quadriceps isometric intermittent fatigue test (QIF test)
Fatigue (VAS) | 16 weeks
  VAS fatigue
Aerobic capacity | 16 weeks
  B-FIT Exercise test
Long function | 16 weeks
  Maximal expiratory pressure (MEP)
Long function | 16 weeks
  Forced vital capacity (FVC)
Long function | 16 weeks
  Maximal inspiratory pressure (MIP)
Balance | 16 weeks
  Mini Balance Evaluation Systems Test (Mini-BESTest)
Pain Questionnaire | 16 weeks
  Brief pain inventory questionnaire
Sleep | 16 weeks
  PROMIS Short Form v1.0 - Sleep Disturbance 8a
Social roles an participation | 16 weeks
  PROMIS Short Form v2.0 - Ability to Participate in Social Roles and Activities 8a
Physical Function | 16 weeks
  PROMIS Short Form v2.0 - Physical Function 20a.
Physical activity | 16 weeks
  Activity tracker

IPD SHARING:
Plan to Share IPD: No